CLINICAL TRIAL: NCT05444959
Title: Evaluation of the Impact of Exercise / Stress Stimuli on the Mechanisms and Efficacy of Beta-hydroxy-beta-methylbutyric Acid (HMB) in Trained and Malnourished Subjects
Brief Title: The Impact of Exercise / Stress Stimuli on HMB Supplementation Efficacy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: National Science Centre, Poland (Other Government); Faculty of Physical Education and Sport at Charles University, Czech Republic (Unknown); Poznan University of Life Sciences, Poland (Unknown); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Prof Dr hab., PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDS2022_0001
Record Dates: First submitted 2022-04-12; First posted 2022-07-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Supplementation; Sport; Sports Nutrition; Sports Dietetics; Protein Kinases; Aerobic Capacity; Fat Free Mass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMB supplementation (Experimental): The experimental procedure for each participant in this group includes a two 21-days periods HMB supplementation.
  HMB will be administered in the form of blinded liquid containing 1 mL HMB free acid per 30 drops. The liquid HMB will be ingested with at least 100 mL of water. Each participant will ingest individualized dose of 90 mg HMB/kgFFM/day of liquid HMB free acid in a split dose per day. On training days in the S group during the first and the second period of supplementation and on training days in W group during the second period of supplementation the supplement will be taken before (half of the individual daily dose) and immediately after training session (second half of the individual daily dose), On rest days the supplements will be taken in the morning (half of the individual daily dose) and before bedtime (second half of the individual daily dose).
  Interventions: Dietary Supplement: HMB supplementation
- Placebo treatment (Placebo Comparator): The experimental procedure for each participant in this group includes a two 21-days periods Placebo supplementation.
  PLA (liquid placebo similar in appearance, taste and smell to HMB, but containing no HMB) will be placed in the blinded liquid form. PLA will be ingested with at least 100 mL of water. Each participant will ingest individualized dose of 90 mg PLA/kgFFM/day of liquid PLA in a split dose per day. On training days in the S group during the first and the second period of supplementation and on training days in W group during the second period of supplementation, the PLA will be taken before (half of the individual daily dose) and immediately after training session (second half of the individual daily dose), On rest days the PLA will be taken in the morning (half of the individual daily dose) and before bedtime (second half of the individual daily dose).
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: HMB supplementation — Group taking oral HMB free acid supplementation in a blinded liquid form.
  Arms: HMB supplementation
Dietary Supplement: Placebo treatment — Group taking oral supplementation with placebo (in a blinded liquid form).
  Arms: Placebo treatment

SUMMARY:
The study aims at assessing the influence of β-hydroxy-β-methylbutyrate (HMB) free acid supplementation (90 mg/kg of fat free body mass/day) supplemented for 21 days on protein kinases activity and selected hormones levels, and subsequent improvements in muscle protein synthesis, lean body mass content and aerobic capacity.

DETAILED DESCRIPTION:
The main aim of the project is to assess the effects of 21 days of HMB (90 mg/kg of fat free body mass per day) or Placebo (PLA) supplementation under two distinct exercise/stress stimulus conditions in the groups of exercise trained participants (S group) and individuals showing features of malnutrition (W group) on the activity of Akt/PBK/mTOR/p70S6K and MAPK/ERK protein kinase pathway in peripheral blood mononuclear cells and muscle; blood concentrations of free and total testosterone, cortisol, IGF-1 and growth hormone; level of resting and exercise energy metabolism rate and alternations in energy sources utilization during exercise, as well as aerobic capacity and body composition.

The study is a double-blind, randomized, placebo-controlled, parallel-group trial. The study protocol consists of two 21-days supplementation periods. Within the first period of the trial the participants will follow their customary physical exercise (S group) / lifestyle (W group). In turn, in the second period of the trial the routine training (S group) or customary lifestyle (W group) will be supplemented twice a week with a functional training program, as a source of an additional exercise/stress stimulus.

Investigators aim to recruit 60 exercise trained individuals (S group) and 60 will be inactive individuals showing features of malnutrition (W group). Random allocation of participants to the HMB and PLA treatments will be done using a random sequence generator, with groups being equalised by fat-free mass level (within S group and W group separately).

At the first preliminary visit anthropometric measurements, and familiarization with exercise test procedures [i.e., incremental cycling test with ergorespirometry, maximal voluntary isometric contraction test (MVIC; performed in a Biodex isokinetic dynamometer)] will be performed. After the completion of the preliminary tests, the participants within S group and W group will be divided randomly into two treatments: 90mg/kgFFM per day of HMB or the same amount of PLA. There will be two 21-days supplementation periods differing in the type of exercise/stress stimulus of the organism.

Before the start of supplementation period (T1) and after their completion (T2 and T3) the series of testing procedures will be performed, each of the series will consist of one day. Each testing series (T1, T2, and T3) will include anthropometric measurements followed by pre-exercise (pre-Ex) blood collection (for the determination of the activity of signaling protein kinases in peripheral blood mononuclear cells; hormone concentrations: free and total testosterone, cortisol, IGF-1 and growth hormone; concentrations of alternative energy sources: ketone bodies <acetoacetate and beta-hydroxybutyrate> and free fatty acids; activity of selected enzymes: lactate dehydrogenase <LDH>, and creatine kinase <CK>; gasometric indices: pH, pCO2, pO2 and electrolytes: Ca2+, Na+, K+, Cl-; concentrations of other biochemical indices: myoglobin, urea, creatinine, glucose, lactate, bilirubins ), the m. vastus lateralis ultrasound and collection of the m. vastus lateralis samples using the percutaneous muscle microbiopsy technique (for the determination of the activity of signaling protein kinases). After the resting pre-Ex procedures, the ICT will be performed. Then the post-exercise (post-Ex) blood sampling and second muscle microbiopsy will be carried out. Finally, at the end of the procedures the MVIC will be assessed.

After collection all the data, comparisons between supplementation treatment conditions (HMB vs PLA) within groups and supplementation periods, as well as comparisons between studied groups (S group vs W group) within supplementation treatment and supplementation period will be performed using T-test for independent variables. Comparisons between supplementation periods within studied groups and supplementation treatment will be performed via T-test for dependent variables. Statistical analysis will be performed using Statistica v. 13.3, StatSoft Polska Sp. z o.o., 2022.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from all participants before the study
* a current medical clearance to practice sports,
* Group S: regular physical activity (> 250 minutes per week), training practice (> 10 years),
* Group W: a subjects characterized by lack of regular physical activity that never were trained in competitive sports and certain features of malnutrition/low physical fitness,

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* serious disease or metabolic problems,
* intake of ergogenic supplements 3 months before the beginning of the study,
* history of anabolic androgenic steroids or drugs use that may interfere with muscle mass control (eg, corticosteroids), or affect physical performance,
* smoking and tobacco use,
* presence of infectious disease in the previous 4 weeks of the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the molecular potential after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  AKTser473, mTORSer2448, p70S7K1Thr389, 4E-BP1Ser65/Thr70, and 4EBP1Thr37/46 kinase activity (optical density)

SECONDARY OUTCOMES:
Changes in the muscle cholesterol and mevalonate content (in the vastus lateralis muscle samples) after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Muscle cholesterol and mevalonate content (units)
Changes in blood concentrations of hormones: free and total testosterone, cortisol, IGF-1, growth hormone after supplementation and exercises-induced stress stimuli on the organism. | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Blood free and total testosterone, cortisol, IGF-1, growth hormone content
Changes in creatine kinase (CK) and lactate dehydrogenase (LDH) activity (IU) in blood after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  CK and LDH activity (IU)
Changes in body mass and body mass composition after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Body mass, fat free mass, fat mass (kg)
Changes in maximal oxygen uptake during the incremental cycling test after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  VO2max level (mL/min)
Changes in total body water content after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Body water content (L)
Changes in other biochemical indices: myoglobin, urea, creatinine, glucose, lactate, bilirubins and electrolytes (Ca2+, Na+, K+, Cl-) after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Blood concentrations of : myoglobin (mmol/L), urea (mmol/L), creatinine (mmol/L), glucose (mmol/L), lactate (mmol/L), bilirubins (mmol/L), and electrolytes [Ca2+, Na+, K+, Cl-] (mmol/L)
Changes in utilization of energy substrates during rest and physical exercise after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Utilization of energy substrates - fats, carbohydrate and protein during rest and exercise (g/min)
Changes in resting and exercise energy expenditures after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Energy expenditure during rest and exercise (kcal/min)
Changes in total daily energy expenditures after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Daily energy expenditure (kcal/day)
Changes in specific exercise performance test Fight Gone Bad after supplementation and exercises-induced stress stimuli on the organism | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Number of repetitions of five different exercise - sumo deadlift high-pulls, wall ball shots, box jumps, push press and rowing on an ergometer in each of three exercise rounds and total number of repetitions of all exercises of all exercise rounds (reps
Changes in the maximum voluntary isometric contraction (MVIC) after supplementation and exercises-induced muscle damage | Day 0 [Baseline (before treatment)] and after 21 days of each two supplementation periods
  Maximum voluntary isometric contraction (MVIC) torque (Nm)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, Prof., PhD, Principal Investigator — Department of Sports Dietetics, Poznan University of Physical Education
Locations (2):
- Department of Physiology and Biochemisty at the Faculty of Physical Education and Sport (Charles University, Prague, Czech Republic), Prague, Prague 6, Czechia
- Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided